CLINICAL TRIAL: NCT03142932
Title: COach2Quit TRIAL: Assessing a Prototype Personal Carbon Monoxide Monitor for Smoking Cessation
Acronym: C2Q
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Maryland Department of Health and Mental Hygiene (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00124820
Record Dates: First submitted 2017-04-28; First posted 2017-05-08 (Actual); Results first posted 2018-11-01 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Smoking; Smoking Cessation
Keywords: smoking
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Monitoring, Physiologic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control (Active Comparator): A certified smoking cessation interventionist (SCI) will deliver standardized smoking cessation counseling using the National Cancer Institute (NCI) 5 A's model.
  Interventions: Behavioral: Cessation counseling
- COach2Quit (Experimental): A certified smoking cessation interventionist (SCI) will deliver standardized smoking cessation counseling using the National Cancer Institute's 5 A's model.
  Participants in the COach2Quit arm will be provided with an individualized carbon monoxide (iCO) monitor along with instructions on the use of the monitor and the COach2Quit application.
  Interventions: Device: Individualized carbon monoxide (iCO) monitor; Other: COach2Quit smartphone application; Behavioral: Cessation counseling

INTERVENTIONS:
Device: Individualized carbon monoxide (iCO) monitor — a personal monitor for a breath test for carbon monoxide (CO)
  Arms: COach2Quit
Other: COach2Quit smartphone application — This smartphone application works in conjunction with the iCO monitor
  Arms: COach2Quit
Behavioral: Cessation counseling — The advice to quit smoking message will follow NCI's 5 A's model for smoking cessation counseling. This is a simple smoking cessation counseling strategy with 5 discrete components: (1) Ask about smoking at every opportunity; (2) Advise the patient to quit smoking; (3) Assess readiness to quit; (4) Assist the patient in quitting; and (5) Arrange follow-up.

SUMMARY:
The objective of this study is to conduct a randomized controlled trial to determine whether the use of the COach2Quit application (app) reduces smoking more than brief advice for smoking cessation. The investigators hypothesize that real time biomarker feedback and messaging support from the COach2Quit app will lead to greater smoking cessation rates than brief anti-smoking advice alone. If effective, the COach2Quit app could be an easily accessible and cost-effective tool to help smokers quit. The findings from this trial could have implications for the delivery of future outpatient smoking cessation programs.

DETAILED DESCRIPTION:
The goal of this randomized controlled trial is to assess the efficacy of the novel COach2Quit smartphone application by determining whether the use of this app reduces smoking more than brief anti-smoking advice alone. This will be a two-arm individually randomized trial and participants who are currently smoking will be assigned 1:1 to either study arm. Smoking behavior will be measured through self-report at baseline, 2-week and 1-month follow up visits. Smoking behavior will also be verified by 2 biomarker measurements: carbon monoxide breath test and urine cotinine, collected at baseline, 2-week and 1-month follow-up visits. In addition, participants will receive weekly follow-up calls. The primary outcome will be smoking cessation at the 1-month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* current, daily smokers
* agree to participate and anticipate to be living in Baltimore for at least 2 months
* own a phone that is compatible with the app
* be willing to set at baseline assessment a quit date within 2 weeks

Exclusion Criteria:

* are suffering from any unstable medical condition precluding the use of the CO monitor (e.g. severe COPD)
* are currently using smokeless tobacco including e-cigarettes
* are currently using nicotine replacement therapy or other smoking cessation treatment
* are pregnant, determined by participant self-report
* have a negative baseline result on both urine cotinine AND CO monitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan E Golub, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

REFERENCES:
- See also: 5 As: Treating Tobacco Use and Dependence — http://www.ahrq.gov/clinic/tobacco/5steps.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through posters advertising the study around the Johns Hopkins Medical Institutions East Baltimore campus, including clinics, inpatient and outpatient facilities, and through participant referrals.
Pre-assignment Details: 160 participants were assessed for eligibility, 58 did not meet inclusion criteria
Groups:
- COach2Quit: A certified smoking cessation interventionist (SCI) will deliver standardized smoking cessation counseling using the National Cancer Institute's 5 A's model.
  Participants in the COach2Quit arm will be provided with an individualized carbon monoxide (iCO) monitor along with instructions on the use of the monitor and the COach2Quit application.
  Individualized carbon monoxide (iCO) monitor: a personal monitor for a breath test for carbon monoxide (CO)
  COach2Quit smartphone application: This smartphone application works in conjunction with the iCO monitor
  Cessation counseling: The advice to quit smoking message will follow NCI's 5 A's model for smoking cessation counseling. This is a simple smoking cessation counseling strategy with 5 discrete components: (1) Ask about smoking at every opportunity; (2) Advise the patient to quit smoking; (3) Assess readiness to quit; (4) Assist the patient in quitting; and (5) Arrange follow-up.
Period: Overall Study
Arm/Group | Control | COach2Quit
Started | 52 | 50
Completed | 50 | 39
Not Completed | 2 | 11
Not completed — Lost to Follow-up | 2 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | COach2Quit | Total
Number analyzed (Participants) | 52 | 50 | 102
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 51 [41 to 55] | 52 [47 to 56] | 52 [45 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 28 | 59
  Male | 21 | 22 | 43
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 10 | 6 | 16
  Black/African American | 39 | 42 | 81
  Mixed Race/Other | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 52 | 50 | 102
Education [Count of Participants; unit: Participants]
  Less than high school | 14 | 20 | 34
  High school or more | 38 | 30 | 68
Employment [Count of Participants; unit: Participants]
  Employed (full/part time) | 13 | 6 | 19
  Unemployed/don't work | 39 | 44 | 83
Cigarettes smoked per day [Median (Inter-Quartile Range); unit: cigarettes] | 10 [9 to 20] | 10 [7 to 20] | 10 [8 to 20]
Quit attempts in past 12 months [Median (Inter-Quartile Range); unit: attempts] | 2 [1 to 2] | 2 [2 to 2] | 2 [1 to 2]
Fagerström Test for Nicotine Dependence [Mean (Standard Deviation); unit: score] — We used the Fagerstrom Test for Nicotine Dependence (FTND) to measure nicotine dependence.
  The measure consists of 6 Questions. Each question has multiple response options out of which one option must be selected. Each option carries a corresponding numerical score. The scores for each question are summed to obtain a total score. The range of possible scores is 1 to 10, with a higher value indicating greater nicotine dependence (worse outcome).
  The interpretation of scores is as follows:
  1-2: low dependence 3-4: low to moderate dependence 5-7: moderate dependence 8+: high dependence
  score | 2.85 (1.51) | 2.54 (1.43) | 2.69 (1.47)

OUTCOME MEASURES:

1. Primary Outcome: Smoking Status Using a Point of Care Test for Measuring Carbon Monoxide (CO)
Description: A point of care test for measuring carbon monoxide (CO) will be conducted via the piCO Smokerlyzer from OPS Medical, designed specifically for smoking cessation programs and tobacco control programs. Carbon monoxide will be measured in an exhaled breath in parts-per-million (ppm). A reading of ≤ 10ppm will indicate abstinence.
Time Frame: baseline
Population: Thirteen participants were lost to follow-up (9 at the 14-day visit and 4 at the 30-day visit) and the sample size for the analysis was 89. There were no significant differences in baseline characteristics between participants lost to follow-up and participants who completed the study.
Measure: Median (Inter-Quartile Range); unit: parts per million
Arm/Group | Control | COach2Quit
Number analyzed (Participants) | 50 | 39
parts per million | 22.0 [14.0 to 30.0] | 23.0 [18.0 to 33.0]

2. Primary Outcome: Smoking Status Using a Point of Care Test for Measuring Carbon Monoxide (CO)
Description: as for outcome 1
Time Frame: 1 month
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: parts per million
Arm/Group | Control | COach2Quit
Number analyzed (Participants) | 50 | 39
parts per million | 18.5 [10.0 to 28.0] | 19.5 [15.0 to 26.0]

3. Primary Outcome: Number of Participants With Color Change for Urine Test for Measuring Cotinine
Description: A point of care urine test for measuring cotinine will also be conducted via the SmokeScreen® test from GFC Diagnostics Ltd. to verify smoking status. A color change to red/orange indicates a positive sample, with a darker color indicating greater nicotine intake.
Time Frame: baseline
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Control | COach2Quit
Number analyzed (Participants) | 50 | 39
participants
  Normal / no change | 1 | 1
  Light | 13 | 2
  Moderate | 11 | 13
  Heavy | 8 | 14
  Very Heavy | 12 | 5
  Missing/could not interpret | 5 | 4

4. Primary Outcome: Number of Participants With Color Change for Urine Test for Measuring Cotinine
Description: as for outcome 3
Time Frame: 1 month
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Control | COach2Quit
Number analyzed (Participants) | 50 | 39
participants
  Normal / no change | 1 | 1
  Light | 6 | 2
  Moderate | 11 | 10
  Heavy | 13 | 12
  Very Heavy | 10 | 5
  Missing/could not interpret | 9 | 9

5. Secondary Outcome: Reasons for Quitting Scale
Description: We used the Reasons for Quitting (RFQ) scale to measure motivation to quit smoking. The scale is used to measure intrinsic and extrinsic motivation for quitting smoking. Each item in the scale is evaluated using a 5-point Likert scale regarding how true the statement is about the participant's motivation to quit smoking (Not at all true, a little bit true, moderately true, quite true, extremely true). Each option takes on a numerical score from 0 (not at all true) to 4 (extremely true). Scores are summed across all items in the scale and divided by the number of items in the scale to obtain the RFQ score. The range of possible scores is 0 to 4. A higher score indicates greater motivation to quit smoking.
Time Frame: baseline
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Control | COach2Quit
Number analyzed (Participants) | 50 | 39
score on a scale | 2.6 [2.4 to 2.8] | 2.6 [2.4 to 2.8]

ADVERSE EVENTS:
Time Frame: 6 months (May - November 2017)
Arm/Group | Control | COach2Quit
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/50
Other Adverse Events (participants affected / at risk) | 0/52 | 0/50

LIMITATIONS AND CAVEATS:
Limitations of the study include small sample size, short follow-up duration and large loss to follow-up. Self-reported measures could be subject to recall bias and social desirability bias. We also did not collect information on substance use.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-15): https://cdn.clinicaltrials.gov/large-docs/32/NCT03142932/Prot_SAP_000.pdf